CLINICAL TRIAL: NCT07259616
Title: Incidence of Cervical Cancer in HPV-positive Women With Low-grade Cytological Abnormalities
Status: Completed | Type: Observational
Sponsor: Gynaecologisch Oncologisch Centrum Zuid (Other)
Collaborators: PALGA foundation (Other); Amphia Hospital (Other); Maastricht University (Other)
Responsible Party: Principal Investigator, Jurgen M.J. Piek, Principal investigator, Gynaecologisch Oncologisch Centrum Zuid
Other Study IDs: GOCZ
Record Dates: First submitted 2025-09-24; First posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Cervical Intraepithelial Neoplasia; Cervix Uteri Cancer; Human Papilloma Virus; Cervix Carcinoma; Cervix; Intraepithelial Neoplasia
Keywords: Human papilloma virus; Cervical cancer; Low-grade cytological abnormalities; Cervical cancer screening; Retrospective cohort study; Five-year incidence
MeSH Terms: conditions — Uterine Cervical Dysplasia; Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort low-grade cytological abnormalities: Women who participated in the population-based cervical cancer screening program in the Netherlands between January 2017 and December 2018 who were HPV positive and with cytology results atypical squamous cells of undetermined significance (ASC-US), atypical glandular cells of endocervical origin (AGC), or low-grade squamous intraepithelial lesion (LSIL) according to the Bethesda system.
- Cohort HPV positive and no cervical abnormalities: Women who participated in the population-based cervical cancer screening program in the Netherlands between January 2017 and December 2018 who were HPV positive and with a stable cytology result negative for intra-epithelial neoplasia according to the Bethesda system.

SUMMARY:
The goal of this observational study is to assess the five-year incidence of histologically confirmed cervical cancer among women who test positive for human papillomavirus (HPV) with low-grade cytological abnormalities, to evaluate whether follow-up intensity could be reduced in women participating in the Dutch population-based cervical cancer screening program who are HPV-positive and have low-grade cytological abnormalities - atypical squamous cells of undetermined significance (ASC-US), atypical glandular cells of endocervical origin (AGC), or low-grade squamous intraepithelial lesions (LSIL).

The main questions it aims to answer are:

What is the five-year risk of developing cervical cancer in HPV-positive women with low-grade cytological abnormalities?

Does the presence of subsequent low-grade cytology affect the five-year risk of cervical cancer in this population?

Researchers will compare the risk of cervical cancer in HPV-positive women with low-grade abnormalities to women with stable negative for intraepithelial lesion or malignancy (NILM) cytology, since women with stable NILM are discharged from further follow-up back to the screening programme. This will help evaluate whether follow-up intensity can be reduced in women with low-grade abnormalities.

ELIGIBILITY:
Inclusion Criteria:

Women who participated in the cervical cancer screening program in the Netherlands between January 2017 and December 2018, who:

* Tested HPV-positive with cytology results categorized as atypical squamous cells of undetermined significance (ASC-US), atypical glandular cells of endocervical origin (AGC), or low-grade squamous intraepithelial lesion (LSIL) according to the Bethesda system, or
* Were HPV-positive and had stable negative for intra-epithelial leasion or malignancy (NILM) cytology after one year.

Exclusion Criteria:

* None

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Women/people who have a cervix.
Study Population: This retrospective cohort study included women who participated in the population-based cervical cancer screening program in the Netherlands between January 2017 and December 2018. Eligible participants were HPV-positive and had cytology results categorized as atypical squamous cells of undetermined significance (ASC-US), atypical glandular cells of endocervical origin (AGC), or low-grade squamous intraepithelial lesion (LSIL) or stable negative for intra-epithelial leasion or malignancy (NILM) cytology results after one year according to the Bethesda system.
Sampling Method: Probability Sample
Enrollment: 46079 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Five-year incidence cervical cancer | From enrollment up to 5 years after.
  Incidence of histologically confirmed cervical cancer within the five-year screening interval.

SECONDARY OUTCOMES:
Time to diagnosis of cervical carcinoma | From enrollment up to 5 years after.
  Time from enrollment to diagnosis of cervical carcinoma
All-cause mortality | From enrollment up to 5 years after.
  The number of participants that died from enrollment up to five years after, all causes of death included.
Examination at which the diagnosis cervical carcinoma was established | Moment of diagnosis of cervical carcinoma from enrollment up to 5 years after.
  Type of examination at which the diagnosis was established
Carcinoma subtype | Moment of diagnosis of cervical carcinoma within 5 years after enrollment.
  Histological characteristics of carcinoma (subtype).
Incidence of cervical cancer within 5 years of inclusion stratified by histological diagnosis within three months of enrollment | From enrollment up to 5 years after.
  Incidence of cervical cancer within 5 years of inclusion stratified by histological diagnosis within three months of baseline abnormal cytology (≤ CIN I vs CIN 2+) and, for the ≤ CIN I group, fur-ther stratified by cytology at 12-month follow-up (no or nondiagnostic cytology, ≤ LSIL, HSIL +).

IPD SHARING:
Plan to Share IPD: No
We do not have ownership of the individual participant data. Data can be obtained on request at https://aanvraag.palga.nl/login

REFERENCES:
- [Background] Cervical cancer screening programme. RIVM n.d. https://www.rivm.nl/en/cervical- cancer-screening-programme (accessed June 1, 2025).
- [Background] WHO guideline for screening and treatment of cervical pre-cancer lesions for cervical cancer prevention [Internet]. 2nd edition. Geneva: World Health Organization; 2021. Available from http://www.ncbi.nlm.nih.gov/books/NBK572317/ PMID 34314129
- [Background] Eramus MC, Palga. Bevolkingsonderzoek Baarmoederhalskanker - Monitor 2017. RIVM 2017.
- [Background] The Netherlands: Integraal Kankercentrum Nederland. National Guidelines: CIN, AIS en VAIN (Dutch). Richtlijnendatabase Federatie Medisch Specialisten;Accessed June 2025.
- [Background] The Netherlands: Integraal Kankercentrum Nederland. National Guidelines: Cervixcytologie- Codering van de uitslag (Dutch). Richtlijnendatabase Federatie Medisch Specialisten; Accessed June 2025.
- [Background] Sharp L, Cotton S, Cruickshank M, Gray NM, Harrild K, Smart L, Walker LG, Little J; TOMBOLA Group. The unintended consequences of cervical screening: distress in women undergoing cytologic surveillance. J Low Genit Tract Dis. 2014 Apr;18(2):142-50. doi: 10.1097/LGT.0b013e31829c97d8. PMID 24270192
- [Background] Katki HA, Gage JC, Schiffman M, Castle PE, Fetterman B, Poitras NE, Lorey T, Cheung LC, Raine-Bennett T, Kinney WK. Follow-up testing after colposcopy: five-year risk of CIN 2+ after a colposcopic diagnosis of CIN 1 or less. J Low Genit Tract Dis. 2013 Apr;17(5 Suppl 1):S69-77. doi: 10.1097/LGT.0b013e31828543b1. PMID 23519308
- [Background] Ciavattini A, Serri M, Di Giuseppe J, Liverani CA, Gardella B, Papiccio M, Delli Carpini G, Morini S, Clemente N, Sopracordevole F. Long-term observational approach in women with histological diagnosis of cervical low-grade squamous intraepithelial lesion: an Italian multicentric retrospective cohort study. BMJ Open. 2019 Jul 3;9(7):e024920. doi: 10.1136/bmjopen-2018-024920. PMID 31272971
- [Background] Bosch FX, Manos MM, Munoz N, Sherman M, Jansen AM, Peto J, Schiffman MH, Moreno V, Kurman R, Shah KV. Prevalence of human papillomavirus in cervical cancer: a worldwide perspective. International biological study on cervical cancer (IBSCC) Study Group. J Natl Cancer Inst. 1995 Jun 7;87(11):796-802. doi: 10.1093/jnci/87.11.796. PMID 7791229
- [Background] Jansen EEL, Zielonke N, Gini A, Anttila A, Segnan N, Voko Z, Ivanus U, McKee M, de Koning HJ, de Kok IMCM; EU-TOPIA consortium. Effect of organised cervical cancer screening on cervical cancer mortality in Europe: a systematic review. Eur J Cancer. 2020 Mar;127:207-223. doi: 10.1016/j.ejca.2019.12.013. Epub 2020 Jan 21. PMID 31980322
- [Background] Melnikow J, Henderson JT, Burda BU, Senger CA, Durbin S, Weyrich MS. Screening for Cervical Cancer With High-Risk Human Papillomavirus Testing: Updated Evidence Report and Systematic Review for the US Preventive Services Task Force. JAMA. 2018 Aug 21;320(7):687-705. doi: 10.1001/jama.2018.10400. PMID 30140883
- [Background] US Preventive Services Task Force; Curry SJ, Krist AH, Owens DK, Barry MJ, Caughey AB, Davidson KW, Doubeni CA, Epling JW Jr, Kemper AR, Kubik M, Landefeld CS, Mangione CM, Phipps MG, Silverstein M, Simon MA, Tseng CW, Wong JB. Screening for Cervical Cancer: US Preventive Services Task Force Recommendation Statement. JAMA. 2018 Aug 21;320(7):674-686. doi: 10.1001/jama.2018.10897. PMID 30140884
- [Background] Bruni L, Serrano B, Roura E, Alemany L, Cowan M, Herrero R, Poljak M, Murillo R, Broutet N, Riley LM, de Sanjose S. Cervical cancer screening programmes and age-specific coverage estimates for 202 countries and territories worldwide: a review and synthetic analysis. Lancet Glob Health. 2022 Aug;10(8):e1115-e1127. doi: 10.1016/S2214-109X(22)00241-8. PMID 35839811
- [Background] Arbyn M, Weiderpass E, Bruni L, de Sanjose S, Saraiya M, Ferlay J, Bray F. Estimates of incidence and mortality of cervical cancer in 2018: a worldwide analysis. Lancet Glob Health. 2020 Feb;8(2):e191-e203. doi: 10.1016/S2214-109X(19)30482-6. Epub 2019 Dec 4. PMID 31812369

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-11-20): https://cdn.clinicaltrials.gov/large-docs/16/NCT07259616/Prot_SAP_000.pdf